CLINICAL TRIAL: NCT00593437
Title: T-score Comparability Between GE Lunar Prodigy and Norland Excel Densitometers
Acronym: Wildwood
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-1053
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2010-04

CONDITIONS: Bone Densitometry
Keywords: bone density diagnostic equipment discrepancies

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: diagnosed with normal bone density by Norland Excel
- 2: diagnosed with osteopenia by Norland Excel densitometer
- 3: diagnosed with osteoporosis by Norland Excel densitometer

SUMMARY:
Differences in determining bone density scores have been found when comparing different bone density machines. Reducing differences between machines will improve diagnostic agreement for patients measured at different clinics. This study will test if this difference exists between the Norland Excel, such as the one at Wildwood Clinic, and the GE Healthcare Lunar Prodigy at the UW Osteoporosis Clinical Research Center.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory women age 40 years and older
* Recent spine and hip DXA at Wildwood clinic in Madison, WI

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ambulatory women age ≥ 40 who have recently had a spine and hip DXA at the Wildwood Clinic on a Norland Excel densitometer
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2006-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Spine and hip BMD and T-score measurements will be compared between densitometry machines. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, MD, Principal Investigator — University of Wisconsin - Institute on Aging
Locations (1):
- University of Wisconsin Osteoporosis Clinical and Research Program, Madison, Wisconsin, United States